CLINICAL TRIAL: NCT03153202
Title: Study to Evaluate the Safety and Preliminary Efficacy of Ibrutinib and Pembrolizumab in Patients With Chronic Lymphocytic Leukemia (CLL) or Mantle Cell Lymphoma (MCL)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joshua Brody (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Joshua Brody, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-0554
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Chronic Lymphocytic Leukemia; Mantle Cell Lymphoma
Keywords: Ibrutinib; Pembrolizumab; Chronic Lymphocytic Leukemia; Mantle Cell Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell | interventions — ibrutinib; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a non-randomized trial. Patients will be allocated to appropriate cohort A-D per their disease type and time of enrollment to study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with CLL (Experimental): Participants with relapsed/ refractory Chronic Lymphocytic Leukemia (CLL) or 17p- CLL
  Interventions: Drug: Ibrutinib; Drug: Pembrolizumab
- Participants with MCL (Experimental): Participants with relapsed/ refractory Mantle Cell Lymphoma (MCL)
  Interventions: Drug: Ibrutinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Ibrutinib — once daily oral intake ibrutinib
Drug: Pembrolizumab — 200mg IV pembrolizumab on Day 1 of each cycle

SUMMARY:
The purpose of this study is to determine the most appropriate dose for the combination of ibrutinib and pembrolizumab and to see if the combination is active for the disease. The study will monitor for any side effects and if the combination of ibrutinib and pembrolizumab works in the cancers being studied.

There will be 2 experimental drugs given to the subject in this study. One experimental drug used in this study is called ibrutinib and the second is called pembrolizumab.

This is the first time that ibrutinib will be used in combination with pembrolizumab. This combination is considered experimental. Experimental means that it is still being tested to see if it is safe and effective. Ibrutinib is a new drug known as a 'Bruton's Tyrosine Kinase (BTK) inhibitor'. Ibrutinib blocks an enzyme (protein) that affects how certain types of blood cancer cells grow and survive. Blocking this enzyme is a very important mechanism in killing blood cancer cells. Ibrutinib has been approved in the United States, Israel, and the European Union for use in adult patients with mantle cell lymphoma (MCL) and adult patients with chronic lymphocytic leukemia (CLL) who have received at least one prior therapy. Pembrolizumab is an antibody (a type of human protein) that is being tested to see if it will allow the body's immune system to work against tumor cells. Pembrolizumab is approved for use by the U.S. Food and Drug Administration (FDA) for the treatment of adult patients with melanoma (skin cancer) who have received prior treatments. Pembrolizumab is not FDA approved to treat patients with chronic lymphocytic leukemia [CLL] and mantle cell lymphoma [MCL].

DETAILED DESCRIPTION:
(1) Objective: a. (Phase 1) Assess the safety of fixed dose or, as needed, de-escalated ibrutinib/pembrolizumab in patients with MCL (Cohort A) and CLL (Cohort B) to determine recommended phase 2 dosing.

b. (Phase 2A): Assess CR rate of combination ibrutinib/pembrolizumab therapy, in comparison to historical data of ibrutinib monotherapy, in patients with MCL (Cohort C) and CLL (Cohort D).

Hypothesis:

This is an open-label Phase 1/2A study, which consists of Phase 1 (Safety Assessment Cohorts) utilizing a 3+3 dose de-escalation design and Phase 2A (Expansion Cohorts) utilizing a single arm one-stage design.

All patients receive a 28 day lead-in of ibrutinib and thereafter, a treatment 'cycle' is defined as a course of treatment of 21 days starting with the intravenous administration of pembrolizumab on Day 1 of each cycle along with once daily oral intake of ibrutinib on all days.

1. The combination of ibrutinib and pembrolizumab will be safe and well tolerated.
2. The combination of ibrutinib and pembrolizumab will result in higher CR rates compared to historic data of ibrutinib monotherapy in cohorts of CLL and MCL.

Secondary Objectives & Hypotheses

(1) Objective: (Phase 2A): Assess duration of response, overall response rate, and duration of stable disease, compared to historical data of single agent ibrutinib, in patients with MCL (Cohort C) and CLL (Cohort D).

Hypothesis: The combination of ibrutinib and pembrolizumab will increase duration of response, overall response rate and duration of stable disease when compared to historical data of single agent ibrutinib.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be ³ 18 years of age on day of signing informed consent.c
3. Have measurable disease based on:

   1. Lugano classification [6] (cohorts A,C)
   2. International Workshop on CLL [7] (cohorts B,D)
4. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen or leukemic blood sample, only upon written agreement from the Study PI.
5. Have a performance status of 0 or 1 on the ECOG Performance Scale.
6. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 14 days of treatment initiation.
7. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

   Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
9. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active Bacillus Tuberculosis (TB)
4. Hypersensitivity to ibrutinib or pembrolizumab or any of their excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or lymphomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include lymphomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 1 year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a systemic treatment.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent. Patients
16. Has previously received a btk inhibitor and had progressive disease during therapy. Patients who have previously discontinued btk inhibitor therapy because of intolerance may be considered for eligibility per the assessment of the PI and treating physician if there is reason that the patient may better tolerate btk inhibitor therapy at enrollment versus previously.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., hepatitis C virus (HCV) RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2017-07-14 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | up to 3 months
  Safety of fixed dose as determined by DLT to determine recommended phase 2 dosing

SECONDARY OUTCOMES:
Complete Response (CR) rate | up to 1 year
  Number of participants with complete response to combination ibrutinib/pembrolizumab therapy in Phase 2
Progression-free Survival Rate | up to 1 year
  Phase 2: Number of participants with progression-free disease
Overall Survival Rate | up to 1 year
  Phase 2: Number of Participants alive at 1 year of combination therapy

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Brody, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No